CLINICAL TRIAL: NCT06589752
Title: Replication of the NefIgArd Trial of Effectiveness and Safety of a Targeted-release Formulation of Budesonide in Patients With Primary IgA Nephropathy
Brief Title: Replication of the NefIgArd Trial of TRF-budesonide in Primary IgAN
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xie Jingyuan, MD, professor, Ruijin Hospital
Other Study IDs: RepIgAN
Record Dates: First submitted 2024-07-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Budesonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Treat: TRF-budesonide enteric-coated capsule（TARPEYO）
  Interventions: Drug: TARPEYO 4 MG Delayed Release Oral Capsule
- Control: RAS blocker
  Interventions: Drug: RAS inhibitor

INTERVENTIONS:
Drug: TARPEYO 4 MG Delayed Release Oral Capsule — TARPEYO dispensing claim for any dose is exposure
  Groups: Treat
Drug: RAS inhibitor — RASi dispensing claim for any dose is reference
  Groups: Control

SUMMARY:
This replication of the NefIgArd trial of TRF-budesonide aims to use real-world data to evaluate the efficiency and safety of TRF-budesonide in the treatment of IgA nephropathy, from completing real-world research to providing real-world evidence.

DETAILED DESCRIPTION:
Currently, TRF-budesonide are the first specific treatment for IgA nephropathy that targets intestinal mucosal immunity. Results from part A of the Phase III clinical trial (NCT03643965) show that compared to the placebo group, the TRF-budesonide group significantly reduced proteinuria and hematuria, stabilized renal function, and lowered circulating Gd-IgA1 levels at 12 months. However, further real-world studies are needed to verify the efficiency and safety of this treatment for IgA nephropathy. Therefore, this replication trial of the part A of the Phase III clinical trial NefIgArd and evaluates the efficiency and safety of TRF-budesonide in treating IgA nephropathy based on existing observational data, aiming to complete real-world research to provide real-world evidence that can guide clinical practice for IgA nephropathy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years;
2. Primary IgA nephropathy confirmed by renal biopsy;
3. Stable use of RAS blockers;
4. 24-hour urine albumin quantitation ≥1g/day, or urine protein/creatinine ratio ≥0.8g/g (≥90 mg/mmol);
5. eGFR ≥30 mL/min/1.73m².

Exclusion Criteria:

1. Systemic diseases that may cause interstitial IgA deposition, including but not limited to anaphylactoid purpura, systemic lupus erythematosus, herpetic dermatitis, and ankylosing spondylitis;
2. Patients who have received kidney transplants;
3. Those with other glomerular diseases (such as C3 glomerular disease or diabetic nephropathy) and nephrotic syndrome;
4. Patients with acute, chronic, or latent infectious diseases, including hepatitis, tuberculosis (TB), human immunodeficiency virus (HIV), and chronic urinary tract infections;
5. Patients with cirrhosis or severe liver function impairment, as assessed by the investigator;
6. Patients diagnosed with poorly controlled type 1 or type 2 diabetes;
7. Patients with a history of unstable angina, grade III or IV congestive heart failure, and/or arrhythmia as assessed by the investigator;
8. Patients with poorly controlled blood pressure with systolic or diastolic blood pressure ≥140mmHg or 90mmHg. At least one blood pressure measurement should be in the above range (based on up to three measurements, 1 minute apart, taken after resting in the supine position for at least 5 minutes);
9. Patients diagnosed with malignancy within the last 5 years, with the exception of treated basal cell carcinoma of the skin, curably resected squamous cell carcinoma of the skin, polyps of the colon, or carcinoma in situ of the cervix;
10. Patients with osteoporosis who are known to be at moderate or high risk. Chinese patients are defined according to the Asian Osteoporosis Self-Assessment Tool (OSTA) Index;
11. Patients with known glaucoma, known history of cataract and/or cataract surgery that may interfere with study drug action or release (such as peptic ulcer disease, inflammatory bowel disease, and chronic diarrhea);
12. Patients who are allergic to budesonide or any component of the investigational drug formulation;
13. Patients who have previously had a severe adverse reaction to steroids;
14. Patients with psychotic symptoms;
15. Have received any systemic glucocorticoid therapy within 3 months prior to medication;
16. Received immunosuppressants or biologics within 3 months prior to medication;
17. Patients taking potent inhibitors of the cytochrome P450 3A4 enzyme (CYP3A4);
18. Current or former (within the last 2 years) alcohol or drug abuse;
19. Patients who are unwilling or unable to meet program requirements;
20. Life expectancy <5 years;
21. Women who are pregnant, nursing, or unwilling to use contraception during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary IgA nephropathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Change in Urinary Protein Levels from Baseline at 9 months Primary endpoint | 9 months
  Assessment of the change in 24-hour urine protein levels from baseline after 9 months of follow-up.
Change in eGFR from Baseline at 9 Months | 9 months
  Measurement of the change in estimated glomerular filtration rate (eGFR) from baseline after 9 months of follow-up.

SECONDARY OUTCOMES:
Change in 24-Hour Urine Protein Levels Compared to Baseline at 12 Months | 12 months
  Assessment of the change in 24-hour urine protein levels from baseline after 12 months of follow-up.
Change in eGFR Compared to Baseline at 12 Months | 12 months
  Measurement of the change in estimated glomerular filtration rate (eGFR) from baseline after 12 months of follow-up.
Incidence Rate of Adverse Events | 12 months
  Calculation of the incidence rate of adverse events during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, China